CLINICAL TRIAL: NCT03895359
Title: A Phase III Randomized Trial of Transarterial Chemoembolization (TACE) Versus TACE Plus Stereotactic Body Radiation Therapy (SBRT) in Primary or Secondary Liver Carcinoma
Brief Title: Transarterial Chemoembolization (TACE) Versus TACE Plus Stereotactic Body Radiation Therapy (SBRT) in Liver Carcinoma
Acronym: TACE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: CancerCare Manitoba (Other)
Responsible Party: Principal Investigator, Michael Lock, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TACE
Record Dates: First submitted 2019-03-21; First posted 2019-03-29 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transarterial Chemoembolization (TACE) (Active Comparator): Transarterial Chemoembolization (TACE)
  Interventions: Drug: Transarterial Chemoembolization
- TACE Plus Stereotactic Body Radiation Therapy (SBRT) (Active Comparator): Stereotactic Body Radiation Therapy (SBRT)
  Interventions: Radiation: Stereotactic Body Radiation

INTERVENTIONS:
Radiation: Stereotactic Body Radiation — For patients randomized to the SMRT arm, SBRT is to be delivered over 5 fractions delivered over 5 to 15 days.
  Arms: TACE Plus Stereotactic Body Radiation Therapy (SBRT)
Drug: Transarterial Chemoembolization — Transarterial chemoembolization is a standard treatment for patients with hepatocellular carcinoma (liver cancer). Chemotherapy is injected into the arteries of the liver and liver cancer.
  Other Names: TACE
  Arms: Transarterial Chemoembolization (TACE)

SUMMARY:
Trans-arterial chemoembolization (TACE) is a standard treatment for patients with hepatocellular carcinoma (also called liver cancer). This is where chemotherapy is injected into the arteries of the liver and liver cancer. Unfortunately, the tumour grows after TACE in many patients.

A new treatment using a specialized radiation procedure called Stereotactic ablative body radiotherapy (SBRT) may increase the chance to control liver cancer. SBRT allows radiation treatments to be focused more precisely, and be delivered more accurately than with older treatments. The purpose of this study is to find out if TACE alone versus TACE plus SBRT is better for you and your liver cancer.

DETAILED DESCRIPTION:
HCC tends to remain within the liver and, therefore, cure with preserved liver function is possible.4 Treatments with relatively high success rates include surgical resection and liver transplantation. Surgical resection results in 5-year survival rates of approximately 60%-70%.4 Liver transplantation can cure both the cancer and underlying liver disease with 4-year survival for HCC within the Milan criteria (single HCC <5 cm or ≤3 HCC <3 cm) at 70%-85% after transplantation.5 Unfortunately, most patients are not resectable due to the extent of disease. Transarterial chemoembolization (TACE) has become the mainstay of treatment for unresectable HCC. 5,6 TACE is relatively safe due to the liver's unique vascular supply from the portal vein. HCC on the other hand, is supplied almost entirely by branches of the hepatic artery.7 In a randomized controlled trial for unresectable HCC not suitable for a curative intent, transarterial chemoembolisation or TACE were compared to conservative treatment.8 TACE induced objective responses (complete and partial response) that were sustained for at least 6 months in 35% of cases. Survival probabilities at 1 year and 2 years were 82% and 63% for TACE, significantly better than 63% and 27% obtained with conservative treatment. Overall survival at 1 and 2 years was also significantly better for the chemoembolization group 57% and 31% vs. 32% and 11%. However, many patients have large tumours and response rates to TACE decline rapidly with increasing size.9 TACE alone resulted in 2 year overall survivals of 42%, 0 and 0 for lesions 5-7cm, 8-10cm, and >10cm, respectively. Therefore, additional locally ablative treatments are being sought. In the same report, TACE plus radiation resulted in 2 year overall survivals of 63%, 50% and 17% for lesions 5-7cm, 8-10cm, and >10cm, respectively.9 External beam radiotherapy has long been considered to have a very limited role in the treatment of liver tumors. This has historically been because minimum dose required for local ablation exceeded the dose that would result in liver toxicity.10,11 The technical development of stereotactic body radiation therapy (SBRT), alone or in combination with TACE, renewed interest in radiation for HCC.12,13 For SBRT, advanced techniques are used to very accurately deliver a high total dose to the target in a small number of daily fractions while avoiding dose delivery to surrounding healthy structures. This research in HCC was done mainly by two groups, in Michigan and Stockholm, who demonstrated that the delivery of high doses of radiation to limited volumes of the liver had promising results in terms of local control and survival with acceptable toxicity.14,15 SBRT is offered as an ablative radical local treatment. In total as of 2015, eleven primary series reported on tumor response and survival of around 300 patients who have been treated with stereotactic body radiation therapy as primary therapy for HCC (Table A). The reported percentage of objective responses defined as complete and partial was ≥64% in 7 of 8 series. Median survival between 11.7 and 32 months has been observed. Toxicity, based on multiple case series trials, indicate that the treatment is considered safe. The most common CTC grade 3-4 toxicity was elevation of liver enzymes. 16-19 For unresectable cases, both TACE and SBRT have been used safely and with good efficacy as separate treatments. Particularly for larger lesions that are more commonly seen in London, the outcome remains suboptimal compared to surgery. Combined treatment case series have shown dramatic results (Table B), but there has not been any randomized trial to compare the value of combining the two modalities. Therefore, a clinical study comparing SBRT and SBRT+TACE will be significant as it addresses a common problem in one of the two most deadly cancers.

ELIGIBILITY:
Inclusion Criteria:

* Primary hepatobiliary cancer confirmed pathologically
* Non - lymphoma liver metastases confirmed pathologically
* Radiographic liver lesions most consistent with metastases, in a patient with known pathologically proven non - lymphoma cancer and a previously negative CT or MRI of the liver
* Hepatocellular carcinoma diagnosed with vascular enhancement of the lesion consistent with hepatocellular carcinoma, and with an elevated AFP, in the setting of cirrhosis or chronic hepatitis.
* ≤ 5 liver lesions measurable on a contrast - enhanced liver CT or MRI performed within 90 days prior to study entry.
* Primary liver lesion or liver metastases measuring ≤ 25 cm.
* Extrahepatic cancer is permitted if liver involvement is judged to be life - limiting.
* All intrahepatic disease must be encompassed within the radiation fields according to protocol criteria.
* Patient must be judged medically or surgically unresectable
* Zubrod Performance Scale = 0 - 3
* Age > 18
* All intrahepatic disease must be amenable to TACE
* Previous liver resection or ablative therapy is permitted.
* Chemotherapy must be completed at least 2 weeks prior to radiation therapy or TACE, and not planned to be administered for at least 1 week (for anthracyclines at least 4 weeks) after completion of treatment.
* Life expectancy > 6 months.
* Women of childbearing potential and male participants must practice adequate contraception.
* Patient must sign study specific informed consent prior to study entry.

Pretreatment Evaluations Required for Eligibility:

* A complete history and general physical examination.
* CBC, INR, Total bilirubin, albumin, alkaline phosphatase, ALT, AST within 4 weeks prior to study entry. Appropriate levels are as follows:
* Absolute neutrophil count (ANC) ≥ 1,500 cells / mm3
* Platelets ≥ 70,000 cells / mm3
* Hemoglobin ≥ 8.0 g / dl (Note: The use of transfusion or other intervention to achieve Hgb ≥ 8.0 g / dl is acceptable.)
* Total bilirubin < 3 mg / dL
* Prothrombin time / INR < 2 (if not on anticoagulants)
* Albumin ≥ 28 g / L
* AST and ALT < 10 times ULN

Exclusion Criteria:

* Severe cirrhosis or liver failure defined as Child Pugh > B7
* Primary liver tumor or liver metastasis > 25 cm in maximal dimension.
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields
* Severe, active co-morbidity, defined as limiting the patients life to less than 6 months
* Active hepatitis or clinically significant liver failure.
* Pregnancy, nursing women, or women of childbearing potential, and men who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the treatment involved in this study may be teratogenic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2019-05-27 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | At 2 years from start of treatment
  Overall Survival-number of patients alive censored for deaths by any cause
Time to Intrahepatic Progression | Pre-treatment, at 1 month and 3 month follow-up, and at follow-up every 3 months up to 2 years
  This will be measured using the modified RECIST (Response evaluation criteria in solid tumors) criteria

SECONDARY OUTCOMES:
Measurement of Response Rate | The sum of the longest diameter (LD) for all target lesions will be calculated and reported as the baseline sum LD. The baseline sum LD will be used as reference by which to characterize the objective tumor.
  Modified RECIST (Response Evaluation Criteria in Solid Tumors) criteria
Local Failure | 5 years
  Within 1 cm from the original tumor volume
Extrahepatic failure | Pre-treatment, at 1 month and 3 month follow-up, and at follow-up every 3 months up to 2 years
  This will be defined as any lesion found to be new or progressing outside the hepatic organ.
Time to intrahepatic progression | Pre-treatment, at 1 month and 3 month follow-up, and at follow-up every 3 months up to 2 years
  This will be measured using the modified RECIST (Response evaluation criteria in solid tumors) criteria
Radiation Therapy Overall Toxicity Assessment | Weekly during treatment, 1 and 3 month follow-up, and every 3 months thereafter up to 2 years
  CTC V4.0 (Common Terminology Criteria version 4.0)
Radiation Therapy Classic Radiation Toxicity Assessment | Weekly during treatment , 1 and 3 month follow-up, and every 3 months thereafter up to 2 years
  Classic RILD (Radiation-induced liver disease)
Radiation Therapy Non-Classic Toxicity Assessment | Weekly during treatment, 1 and 3 month follow-up, and every 3 months thereafter up to 2 years
  Non-classic RILD (Radiation-induced liver disease)
Radiation Therapy Toxicity Assessment | Patients will be assessed at least once during radiation therapy for toxicity
  Measured using Child-Pugh score to indicate the severity of toxicity. Five variables are considered: presence of ascites, encephalopathy, serum levels of albumin, total bilirubin and prolongation of the clotting time. Each of these variables is assigned a score between 1 and 3 according to its severity or degree of abnormality. The sum of the five scores is used to assign a "Child-Pugh grade" of A, B or C to the patient's clinical condition at that point in time. Grade A indicates a well-functioning liver, Grade B indicates significant functional compromise, Grade C indicates decompensation of the liver.
Change in Health related Quality of Life (QOL) | Pre-Treatment, weekly during treatment, 1 and 3 month follow-up, and every 3 months thereafter
  Measured using the EORTC (European Organisation for Research and Treatment of Cancer) QLQ H&N35 (Quality of Life Questionnaire Head & Neck). According to the EORTC scoring guidelines All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
Overall Quality of Life (QOL) | Pre-Treatment, weekly during treatment, 1 and 3 month follow-up, and every 3 months thereafter up to 2 years
  QLQC30 (Quality of Life Questionnaire version 3)
Liver Related Quality of Life (QOL) | Pre-Treatment, weekly during treatment, 1 and 3 month follow-up, and every 3 months thereafter up to 2 years
  FACT-L (Functional Assessment of Cancer Therapy-Lung)
Cost-benefit | Through study completion, an average of 2 years
  A cost benefit analysis will be used to evaluate the total anticipated cost of the project and compare it to the total expected benefits.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lock, M.D., Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- London Health Sciences Centre, London Regional Cancer Program, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No